CLINICAL TRIAL: NCT00385515
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled Study to Evaluate the Efficacy of SNX-1012 in Reducing the Duration and Severity of Ulcerative Oral Mucositis in Patients Receiving Cytotoxic Chemotherapy for Breast or Lung Cancer
Brief Title: Efficacy of SNX-1012 in the Treatment of Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mucosal Therapeutics (Industry)
Responsible Party: Marna Doucette, Coserics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNX-1012-CLN2-006
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Results first posted 2009-03-18 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-04

CONDITIONS: Stomatitis; Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — meclocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SNX-1012 (meclocyline sulfosalicylate) tablets dissolved in water for oral swish and expectorate; 30 mg 4 times daily for 10 days
  Interventions: Drug: SNX-1012 (meclocycline sulfosalicylate)
- 2 (Placebo Comparator): placebo (matched to SNX-1012) tablets dissolved in water for oral swish and expectorate; 4 times daily for 10 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SNX-1012 (meclocycline sulfosalicylate) — tablets to be dissolved in water for oral swish and expectorate; 30 mg, 4 times daily for 10 days
  Arms: 1
Drug: placebo — Tablets to be dissolved in water for oral swish and expectorate; placebo, 4 times daily for 10 days
  Arms: 2

SUMMARY:
Oral mucositis (OM) is a common and debilitating toxicity induced by many chemotherapy (CT) regimens and by radiation to the head and neck. The purpose of this study is to determine the effectiveness of SNX-1012 in decreasing the duration of Grade 2, 3, or 4 oral mucositis (OM) according to World Health Organization (WHO) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Naive to focal radiation therapy in the head and neck regions for cancer prior to CT Cycle 1. Subjects with prior or concomitant radiation therapy to areas other than the head and neck may be enrolled.
* Histologically confirmed diagnosis of breast or lung cancer (NSCLC or SCLC)
* Chemotherapy regimen containing AC ± T or EC ± T (for breast cancer), cisplatin or carboplatin (for NSCLC or SCLC), or doxorubicin (for SCLC)
* Subjects will receive the same regimen and dose of CT in the OM Treatment CT Cycle as was administered in the immediately preceding CT Cycle.
* Subjects will have had OM of WHO Grade of greater than or equal to 2 during CT Cycle 1 or Cycle 2
* Subjects 18 years and older
* Karnofsky Performance Score >=60
* Baseline laboratory assessments:

Hemoglobin (Hgb) level >= 9 g/dL Absolute neutrophil count (ANC) >= 1.5 x 10 to the 9/L Platelet count >= 100 x 10 to the 9/L Serum bilirubin level <= 1.5 times institutional upper limit of normal (ULN) Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) level <= 2 times above ULN

* Females of childbearing potential must have a negative serum or urine pregnancy test result at the screening visit prior to the start of Cycle 1 and at the visit scheduled for <= 48 hours prior to the start of the OM Treatment CT Cycle
* Subjects with reproductive capability must agree to practice adequate contraception methods (males must use condoms or be surgically sterilized; females must be surgically sterilized, post-menopausal for at least 1 year, or use an appropriate double barrier method, prescribed birth control oral contraceptive, patch, implant, or injection during the course of the study and for up to 30 days after completion of study assessments)
* Absence of other serious concurrent medical illness
* Psychologically able to participate and comply with study requirements

Exclusion Criteria:

* Prior history of oral mucositis with previous chemotherapy treatment
* Previous treatment with an anthracycline agent (other than low-dose neoadjuvant therapy)
* Active liver disease or serum AST and/or ALT level > 2 times above ULN
* Currently receiving an investigational agent, planning to receive an investigational agent during the study period, or received an investigational agent within 30 days of the first dose of SNX-1012
* Use of an immunosuppressive regimen of systemic corticosteroids
* Unwilling/unable to receive periodic oral assessments by a study evaluator or unable to complete the daily self-reported outcome questionnaire
* Pregnant or breast-feeding women
* Bronchoalveolar carcinoma
* Metastases to the central nervous system
* Prior or planned focal radiation therapy in the head or neck regions for the treatment of cancer (prior radiation to areas other than the head and neck is permitted)
* Presence of active or history of chronic oral mucosal disease
* Presence or history of any other primary malignancy (curatively treated nonmelanoma skin cancer is allowed)
* History of chronic liver disease
* Active hepatitis A or B
* Unable to receive CT during the OM Treatment CT Cycle at the same regimen and/or dose as in the immediately preceding CT cycle.
* Known sensitivity to tetracyclines
* Known to be seropositive for HIV or HCV
* Use of an immunosuppressive regimen of systemic corticosteroids.
* Current alcohol dependence or drug abuse
* Psychological, social or familial or geographical reasons that would hinder or prevent study visits
* Compromised ability to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (9):
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Florida Research Cancer Institute, Davie, Florida
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Cancer Specialists of South Texas, Corpus Christi, Texas
  - Cancer Outreach Associates, Abingdon, Virginia
  - Morgantown Internal Medicine Group, Morgantown, West Virginia
- India (18):
  - Vedanta Institute of Medical Sciences, Navrangpura, Ahmedabad, Gujarat
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Post Box No. 32, Idgah Hills, Bhopal, Madhya Pradesh
  - Apollo Speciality Hospital, 320, Mount Road, Teynampet, Chennai, Tamil Nadu
  - Dharamshila Cancer Hospital and Research Centre,, Dharamshila Marg, Vasundhara Enclave, Dehli
  - Apollo Hospitals, Jubilee Hills, Hyderabad, Andhra Pradesh
  - Nizams Institute of Medical Sciences, Punjagutta, Hyderabad, Andhra Pradesh
  - Bhagwan Mahavir Cancer Hospital and Research Centre,, Jawaharlal Nehru Marg, Jaipur, Rajasthan
  - S.K Sony Hospital, Vidyadhar Nagar,, Sector-5 Sikar Road, Jaipur, Rajasthan
  - Netaji Subhash Chandra Bose Cancer Hospital & Research Institute, 16A Park Lane, Kolkatta, West Bengal
  - Chittaranjan National Cancer Institute, 37, S.P. Mukherjee Rd., Kolkatta, West Bengal
  - Dayanand Medical College & Hospital, Tagore Nagar, Civil Lines, Ludhiana, Punjab
  - Jaslok Hospital & Research Centre, 15-Dr. G. Deshmukh Marg, Mumbai, Maharashtra
  - Jehangir Hospital,, 32 Sassoon Road, Pune, Maharashtra
  - Ruby Hall Clinic,, 40, Sassoon Road, Pune, Maharashtra
  - Seth Ramdas Shah Memorial Hospital & Research Centre, Fp-402, Gokhle Nagar Road, Shivaji Nagar, Pune, Maharashtra
  - North Bengal Oncology Centre,, Pradhan Nagar, Siliguri, Dist- Darjeeling, West Bengal
  - Regional Cancer Centre, Medical College Campus, Post Bag No. 2417, Trivandrum, Kerala
  - Christian Medical College & Hospital, IDA Scuddar Road, Vellore, Tamil Nadu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 533 subjects were screened during a chemotherapy cycle and those that developed ulcerative oral mucositis and fully recovered were randomized to treatment with study drug during the next chemotherapy cycle
Groups:
- SNX-1012: SNX-1012 (meclocycline sulfosalicylate) tablets dissolved in water for oral swish and expectorate; 30 mg, 4 times daily for 10 days
- Placebo: Placebo tablets (matched to SNX-1012) dissolved in water for oral swish and expectorate; 4 times daily for 10 days
Period: Overall Study
Arm/Group | SNX-1012 | Placebo
Started | 57 | 24
Completed | 53 | 21
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SNX-1012 | Placebo | Total
Number analyzed (Participants) | 57 | 24 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 18 | 66
  >=65 years | 9 | 6 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.9) | 54.5 (12.0) | 52.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 24 | 77
  Male | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 39 | 17 | 56
  India | 18 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Duration of Ulcerative Oral Mucositis
Description: All randomized subjects were directly observed by trained evaluators for at least 10 consecutive days during the chemotherapy cycle to document the duration for those that developed recurrent ulcerative oral mucositis
Time Frame: At least 10 consecutive days beginning on Day 1 of a chemotherapy cycle
Population: Analysis only includes subjects randomized to the 30mg dose of SNX-1012
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SNX-1012 | Placebo
Number analyzed (Participants) | 44 | 21
Days | 2.3 (3.04) | 3.2 (4.68)

2. Secondary Outcome: Number of Participants With Ulcerative Oral Mucositis
Description: All randomized subjects were directly observed by trained evaluators for at least 10 consecutive days during the chemotherapy cycle to identify recurrence of ulcerative oral mucositis.
Time Frame: At least 10 consecutive days beginning on Day 1 of a chemotherapy cycle
Measure: Number; unit: Participants
Arm/Group | SNX-1012 | Placebo
Number analyzed (Participants) | 44 | 21
Participants | 22 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators are restricted from disclosure of results until 24 months after the completion of the Study at all participating research centers. Sponsor can review results communication prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days.